CLINICAL TRIAL: NCT06070376
Title: Comparative Study Between Fully Covered Esophageal Prosthesis (FC-SEMS) and Partially Covered Esophageal Prosthesis (PC-SEMS) in the Palliation of Dysphagia Due to Malignant Neoplasm of Esophagus.
Brief Title: Comparative Study Between (FC-SEMS) and (PC-SEMS) in the Palliation of Dysphagia Due to Malignant Neoplasm of Esophagus.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Principal Investigator, Fauze Maluf Filho, MD, PhD, FASGE, Instituto do Cancer do Estado de São Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NP3080/22
Record Dates: First submitted 2023-09-27; First posted 2023-10-06 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Esophageal Neoplasms; Dysphagia
Keywords: Esophageal Neoplasms; Palliation of dysphagia; Esophageal stent
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): placement of the esophageal prostheses fully covered in the palliative treatment of malignant esophageal obstructions.
  Interventions: Device: Fully Covered Esophageal Prosthesis (FC-SEMS)
- Group B (Active Comparator): placement of the partially covered esophageal prostheses in the palliative treatment of malignant esophageal obstructions.
  Interventions: Device: Partially Covered Esophageal Prosthesis (PC-SEMS)

INTERVENTIONS:
Device: Fully Covered Esophageal Prosthesis (FC-SEMS) — The placement of the Fully Covered Esophageal Prosthesis (FC-SEMS) will be performed under sedation or general anesthesia supervised by the anesthesiologist at the endoscopy service of the Cancer Institute of the State of São Paulo (ICESP). The tests will be performed under radioscopic control. The tests will be performed on an outpatient basis, and hospitalization may occur in case of clinical need.
  Arms: Group A
Device: Partially Covered Esophageal Prosthesis (PC-SEMS) — The placement of the Partially Covered Esophageal Prosthesis (PC-SEMS) will be performed under sedation or general anesthesia supervised by the anesthesiologist at the endoscopy service of the Cancer Institute of the State of São Paulo (ICESP). The tests will be performed under radioscopic control. The tests will be performed on an outpatient basis, and hospitalization may occur in case of clinical need.
  Arms: Group B

SUMMARY:
Esophageal cancer is the seventh most common type of cancer in the world, with an estimated global incidence of 604,100 new cases per year. The main symptom of esophageal cancer is dysphagia, associated or not with weight loss. Unfortunately, due to asymptomatic presentation in the early stages, more than half of patients are diagnosed in advanced stages of the disease, becoming ineligible for treatment with curative intent. In this sense, chemotherapy and radiotherapy are the pillars of palliative treatment, often regressing the injury and improving symptoms. However, some patients persist with dysphagia. In this scenario, esophageal prostheses are one of the main tools in the palliative treatment of esophageal cancer dysphagia, obtaining rapid and lasting relief of dysphagia. This study aims to compare fully covered (FC-SEMS) and partially covered (PC-SEMS) esophageal prostheses in this context, evaluating the number of reinterventions in each group, as well as the occurrence of adverse events. However, it is expected that with the data obtained it is possible to develop clearer and more effective protocols in the palliation of malignant dysphagia of esophageal stenosis.

DETAILED DESCRIPTION:
STUDY DESIGN: Prospective and randomized study will be conducted.

PREPARATION AND TECHNICAL STEPS OF THE PROCEDURE: The placement of the esophageal prosthesis will be performed under sedation or general anesthesia supervised by the anesthesiologist at the endoscopy service of the Cancer Institute of the State of São Paulo (ICESP). The tests will be performed under radioscopic control. The tests will be performed on an outpatient basis, and hospitalization may occur in case of clinical need.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced malignant neoplasm of the esophagus, whether or not undergoing chemotherapy or radiotherapy;
* Dysphagia score greater than 2 or presence of malignant esophagorespiratory fistula;
* Indication of palliation of dysphagia through the placement of esophageal prostheses in a multidisciplinary meeting.

Exclusion Criteria:

* Patients under 18 years;
* Extraesophageal neoplasms;
* Lesions with longitudinal extension less than 30 mm;
* Previous treatment with esophageal prosthesis;
* Tumors easily transposed to standard endoscope (9.8mm).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2023-06-26 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-08-26 (Estimated)

PRIMARY OUTCOMES:
Reinterventions | 2 years
  Number of reinterventions after the procedure.

SECONDARY OUTCOMES:
Adverse events and patency time of the prostheses | 2 years
  Number of adverse events
Patency time of the prostheses. | 2 years
  Days without need a new prothesis or procedure

CONTACTS AND LOCATIONS:
Overall Officials: Fauze Maluf-Filho, PhD, Principal Investigator — Cancer Institute of the state of São Paulo (ICESP)
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, São Paulo, Brazil